CLINICAL TRIAL: NCT05655897
Title: A Prospective, Multicentric Clinical Trial Protocol to Evaluate the Safety and Efficacy of the GeminiOne Transcatheter Valve Edge-to-Edge Repair System for the Treatment of Moderate-severe or Severe Degenerative Mitral Regurgitation With Single-arm Objective Performance Criteria
Brief Title: Safety and Efficacy of the GeminiOne Transcatheter Valve Edge-to-Edge Repair System in Patients With Moderate-severe or Severe Degenerative Mitral Regurgitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peijia Medical Technology (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22CSP001
Record Dates: First submitted 2022-11-30; First posted 2022-12-19 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Mitral Regurgitation; Degenerative Mitral Valve Disease
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A single set of test (Experimental): The GeminiOne Transcatheter Valve Edge-to-Edge Repair System consists of a transcatheter valve clamping system and an adjustable curved introducer catheter.
  Interventions: Device: GeminiOne Transcatheter Valve Edge-to-Edge Repair System

INTERVENTIONS:
Device: GeminiOne Transcatheter Valve Edge-to-Edge Repair System — The transcatheter valve clamp system consists of a valve clamp, an adjustable bend mid-tube, and a manipulated inner tube. The adjustable bend introducer catheter consists of an adjustable bend outer tube and dilator. The valve clip is composed of nickel-titanium alloy, cobalt-chromium-nickel-molybdenum-iron alloy, and polyethylene terephthalate material and contains a closure clip, gripping tab, central mechanism, braid, and suture. The adjustable bend guiding catheter is used to provide access to the transcatheter valve clamping system and to reach the designated position. The adjustable curved mid-tube and manipulated inner tube are used to enable the delivery, gripping, and release process of the valve clips within the body.

SUMMARY:
To observe and evaluate the safety and efficacy of the GeminiOne Transcatheter Valve Edge-to-Edge Repair System in Patients With Moderate-severe or Severe Degenerative Mitral Regurgitation through a prospective, multicenter clinical trial using objective performance criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who volunteer to participate and sign an informed consent form, understand the purpose of the clinical trial and are able to cooperate throughout the trial process;
2. An age ≥ 18 years;
3. Diagnostic transthoracic echocardiogram (TTE) obtained within 90 days and transesophageal echocardiogram (TEE) obtained within 180 days to determine the presence of symptomatic moderate-severe or severe degenerative mitral regurgitation (defined as mitral regurgitation grade ≥3+);
4. Patients' New York Heart Association (NYHA) cardiac function classification (see Appendix II) in grades II, III, or non-ambulatory grade IV；
5. Patients' left ventricular ejection fraction LVEF ≥ 20%;
6. Patients considered to be at high surgical risk by the multidisciplinary cardiac team ;
7. Patients are anatomically suitable for mitral valve repair and suitable for the device under this study as assessed by the multidisciplinary cardiac team;

Elements include, however, are not constrained to the following:

1. Mitral valve orifice area ≥ 4.0 cm2;
2. Left ventricular end-systolic dimension (LVESD) ≤ 60 mm;
3. The primary regurgitant bundle is a non-conjunctive regurgitant bundle and if the secondary regurgitant bundle is present, must be clinically insignificant;
4. Transeptal puncture and femoral venipuncture are feasible; The recommended reference criteria for high surgical risk are: an STS score of ≥8 for surgical valve replacement (see Appendix III) or an STS score of ≥6 for surgical valve repair, or the existence of other high-risk factors, such as the presence of other high-risk elements such as the presence of ≥ 2 warning signs of moderate-severe frailty or the presence of feasible surgical operative limitations or the presence of ≥ 2 main organs dysfunctions that cannot be elevated postoperatively or other surgical high-risk factors that are genuinely existing in the judgment of the independent cardiac surgeon in this study.

Exclusion Criteria:

1. The presence of intra-cardiac space occupancy, thrombus, or bulky organisms as indicated by echocardiography;
2. The presence of other severe heart valve diseases requiring surgical intervention;
3. Leaflet anatomy that may prevent implantation of the valve clip, proper positioning on the leaflet, or prevent adequate reduction of mitral regurgitation by the valve clip. The assessment is based on transesophageal echocardiographic (TEE) mitral valve evaluation within 180 days prior to the subject's registration and includes:

   1. inability of the valve clips to hold sufficient active leaflets;
   2. lack of primary and secondary tendon support in the clamping area;
   3. significant evidence of calcification in the clamping area;
   4. significant fissures in the clamping area;
4. Active endocarditis, pericarditis, or rheumatic heart disease; or mitral valve leaflet changes resulting from endocarditis or rheumatic heart disease;
5. Severe right ventricular insufficiency (e.g. with symptoms of bilateral lower limb edema with increased jugular venous pressure and hepatomegaly); or pulmonary hypertension (pulmonary artery systolic pressure PASA > 70 mmHg as measured by echocardiography);
6. Patients who have had an acute coronary syndrome within 4 weeks, or untreated severe coronary artery stenosis requiring revascularization;
7. Patients with any cardiovascular intervention, cardiac surgery, cardiac resynchronization therapy (CRT, CRT-D), implantation of a buried cardioverter-defibrillator (ICD), etc. within 30 days; or have planned one of these procedures;
8. Patients underwent mitral valve surgery or mitral transcatheter valve surgery before, or have a left atrial appendage occluder device inside；
9. Patients with end-stage heart failure (ACC/AHA stage D), or after cardiac transplantation, or awaiting cardiac transplantation;
10. Patients who are hemodynamically unstable, defined as systolic blood pressure <90 mmHg without postload-reducing drugs, or in cardiogenic shock; or are requiring intra-aortic balloon counterpulsation, or other hemodynamic support drugs or devices;
11. Patients requiring emergency or urgent surgery for any reason;
12. Patients' femoral vein cannot accommodate a 22F catheter or overlaying ipsilateral deep venous thrombosis, as assessed by the investigator, or are anatomically unsuitable for atrial septum puncture; [13
13. Patients with active infection requiring concurrent antibiotic treatment; in the case of temporary disease, antibiotics must be discontinued for at least 14 days before enrollment;
14. Patients with a history of any cerebrovascular accident within 30 days; or a severe symptomatic carotid stenosis (carotid ultrasound suggesting >70% stenosis);
15. Modified Rankin Scale score ≥ 4 (see Annex IV);
16. Patients with a history of acute peptic ulcer or gastrointestinal bleeding within 3 months;
17. Patients with hematological cachexia, including granulocytopenia (WBC <3 x 109/L), anemia (HB < 90 g/L), thrombocytopenia (PLT <50 x 109/L), bleeding disorders, and coagulopathy; or the presence of contraindications to antiplatelet or anticoagulant medication;
18. Patients with a contraindication to transesophageal echocardiography; or a contraindication to general anesthesia；
19. Patients with severe chronic obstructive pulmonary disease (COPD) requiring long-term steroids or continuous home oxygen therapy；
20. Patients with severe hepatic or renal insufficiency (ALT, AST, creatinine > 2 times the upper limit of normal values)；
21. Pregnant or lactating women, or those with a birth plan within 12 months；
22. Patients with known hypersensitivity to device components or contrast media；
23. Patients enrolled in another clinical study and within the follow-up period；
24. Patients with a disease that would make the evaluation of treatment difficult (e.g. cancer, infection, severe metabolic disease, psychiatric disease, etc.); or patients with a life expectancy shorter than 12 months；
25. Patients whose compliance is assessed by the investigator to be poor and are unable to comply with the follow-up schedule and complete the examination; or other situations in which the investigator considers the issue to be unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-11-24 (Actual); Primary Completion 2025-11-24 (Estimated); Study Completion 2029-11-24 (Estimated)

PRIMARY OUTCOMES:
Treatment success | 12 months
  Percentage of patients freedom from: death, surgery for valve dysfunction, and MR > 2+ (moderate to severe (3+) or severe (4+) mitral regurgitation) .

SECONDARY OUTCOMES:
Acute procedural success | Immediately after procedure, Discharge: 1 day after the patient's exit from the cardiac catheterization laboratory
  Successful in GeminiOne implantation, and residual MR of 2+ or less at discharge. An echocardiography echocardiogram at 30 days can be accepted if the discharge image is not available or hard to interpret. A death before discharge or a re-operation of the mitral valve prior to 30 days is defined as acute procedure failure.
Acute device success | Immediately after procedure
  Rate of successful delivery and release of one or more GeminiOne devices with echocardiographic confirmation of leaflet clamping and successful withdrawal of the delivery catheter
Composite of function and re-operation measures | 30 days, 6 months, and 12 months
  Number of patients freedom from postoperative surgery for mitral valve dysfunction.
Cardiac function change | 30 days, 6 months, 12 months, 2 years, 3 years, 4 years and 5 years
  Number of patients with New York Heart Association (NYHA) Function Class I or II.
Quality of life improvement | 12 months
  Change in quality of life (QoL) at 12 months over baseline, as measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ).

OTHER OUTCOMES:
Incidence of major adverse events (MAEs) | 30 days, 6 months, and 12 months
  MAE is defined as a combined clinical endpoint of death, stroke, myocardial infarction, renal failure, and nonelective cardiovascular surgery for device or procedure-related adverse events occurring after transseptal catheterization.
All-cause mortality | 30 days, 6 months, and 12 months
  The percentage of all-cause death includes cardiac death, non-cardiac death, and death from unknown causes.
Cardiac mortality | 30 days, 6 months, and 12 months
  The percentage of cardiac death

CONTACTS AND LOCATIONS:
Locations (1):
- Peiga Medical Technology (Suzhou) Co., Suzhou, Jiangsu, China